CLINICAL TRIAL: NCT03759210
Title: Outcome After Out of Hospital Cardiac Arrest in Bern, Switzerland
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01488
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Resuscitation; Outcome, Fatal; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sudden cardiac arrests is one of the most frequent causes of death. In Switzerland every year 8000-10.000 people suffer from a cardiac arrest. The EuReCa ONE Study showed regional differences in incidence and chances of survival after cardiac arrests in Europe. The current European Resuscitation Council (ERC) resuscitation guidelines 2015 recommend extracorporeal membrane oxygenation (ECMO) as treatment option for therapy refractory out-of-hospital cardiac arrests (OHCA). ECMO used under cardiopulmonary resuscitation (CPR) is called eCPR (extracorporeal CPR). In the year 2018 eCPR is started to be used in Bern, Switzerland. This study investigates retrospectively the survival and neurologic outcome of patients after OHCA in the region of Bern, Switzerland from 2015-2018. The data will be used as baseline for a prospective evaluation of eCPR cases.

The prospective Evaluation of e CPR will last from 2018 - 2022.

ELIGIBILITY:
Inclusion Criteria:

* All OHCA in the region of Bern, Switzerland in the year 2015-2017

Exclusion Criteria:

* if patient has previously declined to be included in a study (advance directive)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All OHCA cases in the region of Bern, Switzerland in the year 2015-2017
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Neurologic Outcome after 30 days | 30 days after OHCA
  CPC 1 - 5 (Cerebral Performance Category Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, Prof., M.D., Study Chair — University Hospital Bern, Bern, Switzerland; Sabine Nabecker, M.D., Principal Investigator — University Hospital Bern, Bern, Switzerland
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebert F, Abt M, Fehr T, Seidl K, Huber M, Ludwig R, Iten M, Greif R, Nabecker S, Fuchs A. Long-term neurological outcome following out-of-hospital cardiac arrest in Switzerland: a single-centre observational study. Front Med (Lausanne). 2026 Jan 2;12:1716369. doi: 10.3389/fmed.2025.1716369. eCollection 2025. PMID 41551516